CLINICAL TRIAL: NCT00954941
Title: Comparative Trial Ondansetron Alone Versus Combination of Ondansetron Plus Aprepitant for Prevention of Nausea and Vomiting With Hematologic Malignancies Receiving Regimens Containing High-dose Cytarabine
Brief Title: Ondansetron Versus Aprepitant Plus Ondansetron for Emesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0615; NCI-2009-01517 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-05

CONDITIONS: Hematologic Diseases; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Chronic Myelogenous Leukemia
Keywords: Hematologic Disorder; Acute myelogenous leukemia; AML; High-risk myelodysplastic syndrome; HR-MDS; Chronic Myelogenous Leukemia; CML; Ondansetron; Zofran; Aprepitant; Emend; L 754030; MK 869; Emesis; Nausea; Vomiting
MeSH Terms: conditions — Hematologic Diseases; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Vomiting; Nausea | interventions — Ondansetron; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Ondansetron (Experimental): Ondansetron 8 mg bolus by vein from 30 minutes before receiving chemotherapy followed by 24 mg by vein continuous infusion daily while receiving chemotherapy until 12 hours after chemotherapy.
  Interventions: Drug: Ondansetron
- Group 2: Ondansetron + Aprepitant (Active Comparator): Ondansetron 8 mg bolus by vein from 30 minutes before receiving chemotherapy followed by 24 mg by vein continuous infusion daily while receiving chemotherapy until 12 hours after chemotherapy. Aprepitant 125 mg capsule by mouth every morning while receiving chemotherapy followed by 80 mg capsule by mouth daily while receiving chemotherapy continued till 1 day after last chemotherapy dose.
  Interventions: Drug: Ondansetron; Drug: Aprepitant

INTERVENTIONS:
Drug: Ondansetron — 8 mg bolus by vein from 30 minutes before receiving chemotherapy followed by 24 mg by vein continuous infusion daily while receiving chemotherapy until 12 hours after chemotherapy.
  Other Names: Zofran
Drug: Aprepitant — 125 mg capsule by mouth every morning while receiving chemotherapy followed by 80 mg capsule by mouth daily while receiving chemotherapy continued till 1 day after last chemotherapy dose.
  Other Names: Emend; L 754030; MK 869
  Arms: Group 2: Ondansetron + Aprepitant

SUMMARY:
The goal of this clinical research study is to compare the effectiveness of receiving a combination of ondansetron and aprepitant to receiving ondansetron alone in helping to prevent nausea and/or vomiting in patients with Acute myeloid leukemia (AML) or high-risk (HR) Myelodysplastic syndromes (MDS) who are receiving cytarabine. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Cytarabine is a drug that is used to treat AML and high-risk MDS. It is known to cause nausea and/or vomiting. All patients that receive cytarabine also receive drugs to help prevent these side effects.

The Study Drugs:

Ondansetron is designed to block the action of serotonin, a substance in the brain that causes chemotherapy-related nausea and vomiting.

Aprepitant is designed to block a different natural substance in the brain that causes chemotherapy-related nausea and vomiting.

Study Groups:

If you are found eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being in either group.

If you are in Group 1, you will receive ondansetron.

If you are in Group 2, you will receive ondansetron and aprepitant.

Study Drug Administration:

Both groups will receive ondansetron by vein from 30 minutes before receiving chemotherapy until 6 to12 hours after chemotherapy. The length of the chemotherapy infusion will be different for all patients.

If you are in Group 2, in addition to ondansetron, you will take 1 capsule of aprepitant every morning while receiving chemotherapy. You will take your last dose of aprepitant the day after your chemotherapy infusion is completed. If you miss a dose of aprepitant, you can take it as soon as you remember.

Study Diary:

You will fill out a study diary every day for the 7 days after the chemotherapy. You will record how often you experience nausea and/or vomiting and any time you need other medications during this study. It should take about 5 minutes to complete each time.

Length of Study:

You will be on study for up to 7 days. You will be taken off study if intolerable side effects occur.

Blood Draws:

Blood (about 1 teaspoon) will be drawn for routine tests after your last dose (+/- 3 days) of study drug.

This is an investigational study. Ondansetron and aprepitant are both FDA approved and commercially available for the prevention of chemotherapy-related nausea and vomiting. Using the drugs in combination is investigational.

Up to 100 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients greater than or equal to 18 years of age.
2. Patients with a diagnosis of acute myelogenous leukemia, high-risk myelodysplastic syndrome, chronic myelogenous leukemia in blast crisis or acute undifferentiated leukemia who will receive chemotherapy with regimens containing high-dose cytarabine (greater or equal 1g/m^2/d for at least 3 days).
3. Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.

Exclusion Criteria:

1. Patients with emesis or grade 2 or 3 nausea present less than or equal to 24 hours before chemotherapy.
2. Patients with ongoing emesis due to any organic etiology
3. Patients with known hypersensitivity to the study drug or to 5-HT3 receptor antagonists
4. Patients receiving pimozide, terfenadine, astemizole, or cisapride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/11/09 to 3/20/2013. All participants registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the 100 participants registered for screening on this study, fifty participants were randomized to Ondansetron alone (Group 1) and forty-eight participants to Ondansetron plus Aprepitant (Group 2).
Period: Overall Study
Arm/Group | Group 1: Ondansetron | Group 2: Ondansetron + Aprepitant
Started | 50 | 48
Completed | 42 | 41
Not Completed | 8 | 7
Not completed — Received treatment at home | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Insurance Denial | 2 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Ineligible | 2 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Registered eligible participants who received one dose of study medication were evaluable for toxicity but had to receive at least five doses to be evaluable for response. Only 90 participants (46 on Group 1 and 44 on Group 2) had one or more doses of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ondansetron | Group 2: Ondansetron + Aprepitant | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Median (Full Range); unit: years] | 56 [30 to 68] | 53 [21 to 70] | 55 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 29 | 26 | 55
Region of Enrollment [Number; unit: participants]
  United States | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Participant Responses
Description: Participant response defined as: Complete response - no emetic episode, no nausea and no rescue medication during the administration of chemotherapy; Partial response - less than or equal to one episode of emesis in 24 hours, no rescue medication, and no more than moderate nausea (grade 2 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)) during chemotherapy. Vomit was defined as expulsion of stomach contents through the mouth, nausea as stomach distress with distaste for food and an urge to vomit, and rescue medication as antiemetic medications given to treat nausea and/or vomit that did not respond to the initial prophylactic regimen. Treatment success was defined as no nausea, no vomiting and no need for rescue medication within the first 6 treatment days with continuous monitoring.
Time Frame: First 6 treatment days
Population: Of the 98 participants in the study, six (6) in Group 1: Ondansetron and nine (9) in Group 2: Ondansetron + Aprepitant were not.evaluable.
Measure: Number; unit: participants
Groups:
- Group 1: Ondansetron: Ondansetron 8 mg bolus by vein from 30 minutes before receiving chemotherapy followed by 24 mg by vein continuous infusion daily while receiving chemotherapy until 12 hours after chemotherapy.
  Ondansetron : 8 mg bolus by vein from 30 minutes before receiving chemotherapy followed by 24 mg by vein continuous infusion daily while receiving chemotherapy until 12 hours after chemotherapy.
- Group 2: Ondansetron + Aprepitant: Ondansetron 8 mg bolus by vein from 30 minutes before receiving chemotherapy followed by 24 mg by vein continuous infusion daily while receiving chemotherapy until 12 hours after chemotherapy. Aprepitant 125 mg capsule by mouth every morning while receiving chemotherapy followed by 80 mg capsule by mouth daily while receiving chemotherapy continued till 1 day after last chemotherapy dose.
  Ondansetron : 8 mg bolus by vein from 30 minutes before receiving chemotherapy followed by 24 mg by vein continuous infusion daily while receiving chemotherapy until 12 hours after chemotherapy.
  Aprepitant : 125 mg capsule by mouth every morning while receiving chemotherapy followed by 80 mg capsule by mouth daily while receiving chemotherapy continued till 1 day after last chemotherapy dose.
Arm/Group | Group 1: Ondansetron | Group 2: Ondansetron + Aprepitant
Number analyzed (Participants) | 42 | 41
participants
  Complete Response | 20 | 21
  Partial Response | 9 | 12
  No Response | 13 | 8

2. Primary Outcome: Treatment Success Rate
Description: Treatment success is defined as no nausea, no vomiting and no need for rescue medication (or complete response) within the first 6 treatment days. Treatment success rate defined as percentage of participants achieving treatment success.
Time Frame: First 6 treatment days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Ondansetron | Group 2: Ondansetron + Aprepitant
Number analyzed (Participants) | 42 | 41
percentage of participants | 48 | 51

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent until 30 days after the last dose of drug. The full study reporting period was three years four months.
Description: Of the 98 participants registered in the study, 90 participants are included in Adverse Event Reporting as evaluable for toxicity having received one dose of treatment medication.
Arm/Group | Group 1: Ondansetron | Group 2: Ondansetron + Aprepitant
Serious Adverse Events (participants affected / at risk) | 3/46 | 3/44
Other Adverse Events (participants affected / at risk) | 43/46 | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ondansetron (N=46) | Group 2: Ondansetron + Aprepitant (N=44)
Death (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ondansetron (N=46) | Group 2: Ondansetron + Aprepitant (N=44)
Pain (General disorders) | 17 (17) | 12 (12)
Abdominal Cramps (General disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anxiety (Nervous system disorders) | 2 (2) | 2 (2)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Brusing (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 17 (17) | 15 (15)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 1 (1)
edema (Blood and lymphatic system disorders) | 4 (4) | 8 (8)
Fatigue (General disorders) | 9 (9) | 12 (12)
Fever (General disorders) | 2 (2) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
headache (General disorders) | 12 (12) | 11 (11)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 6 (6)
Insomnia (General disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jaundice (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Leg Cramps (General disorders) | 1 (1) | 0 (0)
Nausa (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nosebleed (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Nasal Congestion (General disorders) | 0 (0) | 1 (1)
Prolonged QTc (Cardiac disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Sore Throat (General disorders) | 1 (1) | 0 (0)
Sweating (General disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Taste Alteration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Numbness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes